CLINICAL TRIAL: NCT02559609
Title: Interventions for Unemployed Hazardous Drinkers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UConn Health (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Carla Rash, Assistant Professor, UConn Health
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 15-041-2; R01AA023502 (NIH)
Record Dates: First submitted 2015-08-24; First posted 2015-09-24 (Estimated); Results first posted 2023-06-22 (Actual); Last update posted 2024-04-23 (Actual); Status verified 2024-04

CONDITIONS: Unemployment; Hazardous Drinking
MeSH Terms: interventions — Ethanol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- job activity contracting (Active Comparator): Standard services plus job activity contracting and alcohol monitoring
  Interventions: Behavioral: Job relelated activity contracting
- reinforcement for negative alcohol samples (Experimental): Standard services plus job activity contracting and alcohol monitoring plus reinforcement for negative breath alcohol recordings
  Interventions: Behavioral: Contingency management for alcohol abstinence; Behavioral: Job relelated activity contracting
- reinforcement for completing activities (Experimental): Standard services plus job activity contracting and alcohol monitoring plus reinforcement for completing job-related activities
  Interventions: Behavioral: Contingency management for completing job related activities; Behavioral: Job relelated activity contracting
- reinforcement for negative alcohol samples & activities (Experimental): Standard services plus job activity contracting and alcohol monitoring plus reinforcement for negative breath alcohol recordings and for completing job-related activities
  Interventions: Behavioral: Contingency management for alcohol abstinence; Behavioral: Contingency management for completing job related activities; Behavioral: Job relelated activity contracting

INTERVENTIONS:
Behavioral: Contingency management for alcohol abstinence — Participants will earn reinforcement (incentives) for each alcohol negative breath test provided (when prompted to submit a test) during the 12-week intervention period.
  Arms: reinforcement for negative alcohol samples; reinforcement for negative alcohol samples & activities
Behavioral: Contingency management for completing job related activities — Participants will earn reinforcement (incentives) for completing specific job-related activities during the 12-week intervention period.
  Arms: reinforcement for completing activities; reinforcement for negative alcohol samples & activities
Behavioral: Job relelated activity contracting — Participants will complete job-related activity contracts each week with the goal of obtaining employment.

SUMMARY:
Despite recent improvements in the US economy, unemployment remains a significant concern, and estimates indicate that one-third of unemployed persons drink at hazardous levels, adversely impacting their health and abilities to find jobs. Reinforcement interventions are highly efficacious in reducing substance use, and they can be applied to increase job-seeking activities as well. In partnership with CT United Labor Agency, this project is designed to reduce hazardous drinking and enhance active participation in job-seeking activities among those with job loss. It will evaluate the independent and combined effects of reinforcing negative breathalyzer samples and job-seeking activities to ascertain the simplest and most cost-effective approach to improving outcomes in this population. Unemployed individuals with hazardous drinking (N = 280) will be randomly assigned to one of four conditions using a 2 x 2 design: standard care, standard care with reinforcement for submitting negative breathalyzer samples, standard care with reinforcement for job-seeking activities, or standard care plus reinforcement for both negative breathalyzer samples and job-seeking activities. Participants in all conditions will receive usual services part of CT United Labor Agency, along with a novel remote breath alcohol monitoring procedure. The study interventions will be in effect for three months, and participants will be followed for one year. Alcohol and other drug use, employment, psychiatric symptoms, and global measures of health will be assessed throughout treatment and follow-up. Reinforcing negative breathalyzer samples is expected to significantly reduce drinking, and reinforcing job-seeking activities is expected to increase re-employment rates and reduce time until job attainment. Reinforcing both negative breathalyzer samples and job-seeking activities is hypothesized to improve outcomes along both domains. The reinforcement interventions may also decrease psychiatric distress and slow progression of physical decline, common among the unemployed. If efficacious and cost-effective, results from this study may stimulate adoption of reinforcement interventions in the context of unemployment services. Reducing the adverse consequences of hazardous drinking and improving job re-entry may have pronounced benefits in a highly vulnerable segment of the US population.

ELIGIBILITY:
Inclusion Criteria:

* age 18-65 years
* not worked for pay in the formal economy for >4 weeks
* willing to participate in a workforce training program and willing to accept either part-time or full-time work
* hazardous alcohol use defined by AUDIT scores >8, a mean of >2 drinks/drinking day or >14 drinks/week in men (>1 drink/drinking day or >7 drinks/week in women) in the past 2 months, or submission of an alcohol positive breathalyzer (>0.02 g/dl) or EtG positive urine sample
* English or Spanish speaking and able to read at 5th grade level
* have a valid photo ID
* willing and able to use study equipment and sign an off-campus property transfer form

Exclusion Criteria:

* have begun receiving unemployment benefits within the past 4 weeks
* worked full- or part-time <3 months in the past 3 years in the formal or informal economy
* physiological alcohol withdrawal symptoms (score >10 on Clinical Institute Withdrawal Assessment for Alcohol-revised)
* physiological withdrawal symptoms from an illicit drug use disorder
* serious untreated psychiatric illness
* in recovery from gambling disorder

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2016-04-19 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-06-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carla J Rash, Ph.D., Principal Investigator — UConn Health
Locations (1):
- United Labor Agency, Middletown, Connecticut, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Group A - Standard Job Activity Contracting and Alcohol Monitoring: Standard services plus job activity contracting and alcohol monitoring
  activity contracting: participants will complete job-related activity contracts each week with the goal of obtaining employment
- Group B - Reinforcement for Negative Alcohol Samples: Standard services plus job activity contracting and alcohol monitoring plus reinforcement for negative breath alcohol recordings
  contingency management for alcohol abstinence: participants will earn chances to win prizes for each negative breath alcohol recording provided
  activity contracting: participants will complete job-related activity contracts each week with the goal of obtaining employment
- Group C - Reinforcement for Completing Job Activities: Standard services plus job activity contracting and alcohol monitoring plus reinforcement for completing job-related activities
  activity contracting: participants will complete job-related activity contracts each week with the goal of obtaining employment
  contingency management for activity completion: participants will earn chances to win prizes for completing specific job-related activities
- Group D - Reinforcement for Negative Alcohol Samples & Job Activities: Standard services plus job activity contracting and alcohol monitoring plus reinforcement for negative breath alcohol recordings and for completing job-related activities
  contingency management for alcohol abstinence: participants will earn chances to win prizes for each negative breath alcohol recording provided
  contingency management for activity completion: participants will earn chances to win prizes for completing specific job-related activities
Period: Overall Study
Arm/Group | Group A - Standard Job Activity Contracting and Alcohol Monitoring | Group B - Reinforcement for Negative Alcohol Samples | Group C - Reinforcement for Completing Job Activities | Group D - Reinforcement for Negative Alcohol Samples & Job Activities
Started | 50 | 65 | 58 | 67
Completed | 50 | 64 | 58 | 67
Not Completed | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group A - Standard Job Activity Contracting and Alcohol Monitoring | Group B - Reinforcement for Negative Alcohol Samples | Group C - Reinforcement for Completing Job Activities | Group D - Reinforcement for Negative Alcohol Samples & Job Activities | Total
Number analyzed (Participants) | 50 | 65 | 58 | 67 | 240
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 50 | 65 | 58 | 67 | 240
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.10 (9.77) | 45.94 (11.34) | 42.38 (10.89) | 46.37 (10.06) | 45.23 (10.63)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 34 | 30 | 35 | 116
  Male | 33 | 31 | 28 | 32 | 124
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 7 | 8 | 10 | 29
  Not Hispanic or Latino | 46 | 58 | 50 | 57 | 211
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 0 | 0 | 2
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 0 | 1
  Black or African American | 29 | 37 | 25 | 36 | 127
  White | 19 | 24 | 31 | 28 | 102
  More than one race | 0 | 2 | 0 | 0 | 2
  Unknown or Not Reported | 0 | 1 | 2 | 3 | 6
Region of Enrollment [Number; unit: participants]
  United States | 50 | 65 | 58 | 67 | 240

OUTCOME MEASURES:

1. Primary Outcome: Longest Duration of Alcohol Abstinence (Samples) (Physiological Measure)
Description: Greatest number of consecutive breath tests submitted on-time (within 1 hour of prompt) and reading alcohol negative (BAL < 0.02)
Time Frame: 12 weeks
Population: N=234 analyzed. n=6 with no data: n=1 Group B withdrawal; n=5 had no samples submitted (n=1 Group A, n=1 Group B, n=1 group D) or none submitted on-time (n=2 Group B).
Measure: Median (Inter-Quartile Range); unit: number of alcohol negative breath tests
Arm/Group | Group A - Standard Job Activity Contracting and Alcohol Monitoring | Group B - Reinforcement for Negative Alcohol Samples | Group C - Reinforcement for Completing Job Activities | Group D - Reinforcement for Negative Alcohol Samples & Job Activities
Number analyzed (Participants) | 49 | 61 | 58 | 66
number of alcohol negative breath tests | 6.0 [3.0 to 14.0] | 11.0 [5.0 to 26.0] | 7.0 [4.0 to 17.3] | 7.5 [5.0 to 18.3]
Statistical Analysis 1: Comparison: Group A - Standard Job Activity Contracting and Alcohol Monitoring vs Group B - Reinforcement for Negative Alcohol Samples vs Group C - Reinforcement for Completing Job Activities vs Group D - Reinforcement for Negative Alcohol Samples & Job Activities; Group A/C (contrast -1) compared to Group B/D (contrast 1) to test Aim 1; Test type: Superiority; p = .028, Wilcoxon (Mann-Whitney)

2. Primary Outcome: Percent Alcohol Negative Breath Tests
Description: Of alcohol breath tests requested, the percentage submitted on-time (within 1-hour of prompt) and reading alcohol-negative (BAL < .02)
Time Frame: 12 weeks
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: percentage of alcohol negative tests
Arm/Group | Group A - Standard Job Activity Contracting and Alcohol Monitoring | Group B - Reinforcement for Negative Alcohol Samples | Group C - Reinforcement for Completing Job Activities | Group D - Reinforcement for Negative Alcohol Samples & Job Activities
Number analyzed (Participants) | 49 | 61 | 58 | 66
percentage of alcohol negative tests | 90.8 [48.9 to 100.0] | 98.1 [78.9 to 100.00] | 91.2 [66.6 to 100.0] | 97.1 [67.0 to 100.0]
Statistical Analysis 1: Comparison: Group A - Standard Job Activity Contracting and Alcohol Monitoring vs Group B - Reinforcement for Negative Alcohol Samples vs Group C - Reinforcement for Completing Job Activities vs Group D - Reinforcement for Negative Alcohol Samples & Job Activities; Group A/C (contrast -1) compared to Group B/D (contrast 1); Test type: Superiority; p = .027, Wilcoxon (Mann-Whitney)

3. Primary Outcome: Percent of Days Worked for Pay (Missing Data Treated as Missing)
Description: The percentage of days of work for pay (in the formal or informal economy), with the number of days of data in the denominator (missing data considered missing)
Time Frame: 12 weeks
Population: N=228, n=12 no score: n=1 Group B withdrawal; n=1 Group D on disability (no working allowed); no data for n= 2 Group A, n=4 Group B, n=1 Group C, n=3 Group D
Measure: Median (Inter-Quartile Range); unit: percentage of days work occurred
Arm/Group | Group A - Standard Job Activity Contracting and Alcohol Monitoring | Group B - Reinforcement for Negative Alcohol Samples | Group C - Reinforcement for Completing Job Activities | Group D - Reinforcement for Negative Alcohol Samples & Job Activities
Number analyzed (Participants) | 48 | 60 | 57 | 63
percentage of days work occurred | 1.79 [0.00 to 22.99] | 4.76 [0.00 to 24.40] | 6.25 [0.00 to 25.77] | 1.33 [0.00 to 26.19]
Statistical Analysis 1: Comparison: Group A - Standard Job Activity Contracting and Alcohol Monitoring vs Group B - Reinforcement for Negative Alcohol Samples vs Group C - Reinforcement for Completing Job Activities vs Group D - Reinforcement for Negative Alcohol Samples & Job Activities; Group A/B (contrast -1) was compared to Group C/D (contrast 1) to test Aim 2; Test type: Superiority; p = .66, ANOVA; df = 1

4. Primary Outcome: Time to First Worked
Description: From study day 1, the number of days until first worked in the formal or informal economy during the 12-week intervention, censored at day 85.
Time Frame: 12 weeks
Population: N=228 analyzed. n=12 no score: n=1 Group B withdrawal; n=1 Group D on disability (no working allowed); no data for n= 2 Group A, n=4 Group B, n=1 Group C, n=3 Group D
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Group A - Standard Job Activity Contracting and Alcohol Monitoring | Group B - Reinforcement for Negative Alcohol Samples | Group C - Reinforcement for Completing Job Activities | Group D - Reinforcement for Negative Alcohol Samples & Job Activities
Number analyzed (Participants) | 48 | 60 | 57 | 63
days | 79.50 [15.00 to 85.0] | 57.00 [24.00 to 85.0] | 63.00 [16.50 to 85.0] | 63.00 [16.00 to 85.0]
Statistical Analysis 1: Comparison: Group A - Standard Job Activity Contracting and Alcohol Monitoring vs Group B - Reinforcement for Negative Alcohol Samples vs Group C - Reinforcement for Completing Job Activities vs Group D - Reinforcement for Negative Alcohol Samples & Job Activities; Group A/B (contrast -1) compared to Group C/D (contrast 1) to test Aim 2; Test type: Superiority; p = .89, Regression, Cox

5. Secondary Outcome: Percent of Days Worked for Pay (84 Day Intervention Period in the Denominator)
Description: The percent of days worked for pay (in the formal or informal economy), with 84 days (intervention period duration; missing treated as not working) in the denominator
Time Frame: 12 weeks
Population: as for outcome 4
Measure: Median (Inter-Quartile Range); unit: percentage of days work occurred
Arm/Group | Group A - Standard Job Activity Contracting and Alcohol Monitoring | Group B - Reinforcement for Negative Alcohol Samples | Group C - Reinforcement for Completing Job Activities | Group D - Reinforcement for Negative Alcohol Samples & Job Activities
Number analyzed (Participants) | 48 | 60 | 57 | 63
percentage of days work occurred | 1.19 [0.00 to 18.15] | 4.17 [0.00 to 22.02] | 4.76 [0.00 to 23.81] | 1.19 [0.00 to 22.62]
Statistical Analysis 1: Comparison: Group A - Standard Job Activity Contracting and Alcohol Monitoring vs Group B - Reinforcement for Negative Alcohol Samples vs Group C - Reinforcement for Completing Job Activities vs Group D - Reinforcement for Negative Alcohol Samples & Job Activities; Group A/B (contrast -1) compared to Group C/D (contrast 1) to test Aim 2; Test type: Superiority; p = .58, ANOVA; df = 1

6. Secondary Outcome: Longest Duration of Alcohol Abstinence (Days) (Physiological Measure)
Description: Greatest number of consecutive days of submitting all breath tests requested on-time and reading alcohol negative
Time Frame: 12 weeks
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Group A - Standard Job Activity Contracting and Alcohol Monitoring | Group B - Reinforcement for Negative Alcohol Samples | Group C - Reinforcement for Completing Job Activities | Group D - Reinforcement for Negative Alcohol Samples & Job Activities
Number analyzed (Participants) | 49 | 61 | 58 | 66
days | 4.0 [2.0 to 10.0] | 9.0 [3.0 to 19.0] | 5.0 [3.0 to 12.3] | 6.0 [3.0 to 13.5]
Statistical Analysis 1: Comparison: Group A - Standard Job Activity Contracting and Alcohol Monitoring vs Group B - Reinforcement for Negative Alcohol Samples vs Group C - Reinforcement for Completing Job Activities vs Group D - Reinforcement for Negative Alcohol Samples & Job Activities; Group A/C (contrast -1) compared to Group B/D (contrast 1) to test Aim 1; Test type: Superiority; p = .024, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | Group A - Standard Job Activity Contracting and Alcohol Monitoring | Group B - Reinforcement for Negative Alcohol Samples | Group C - Reinforcement for Completing Job Activities | Group D - Reinforcement for Negative Alcohol Samples & Job Activities
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/65 | 1/58 | 0/67
Serious Adverse Events (participants affected / at risk) | 6/50 | 8/65 | 9/58 | 9/67
Other Adverse Events (participants affected / at risk) | 5/50 | 5/65 | 1/58 | 6/67
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A - Standard Job Activity Contracting and Alcohol Monitoring (N=50) | Group B - Reinforcement for Negative Alcohol Samples (N=65) | Group C - Reinforcement for Completing Job Activities (N=58) | Group D - Reinforcement for Negative Alcohol Samples & Job Activities (N=67)
Inpatient substance use treatment (General disorders) | 3 (5) | 3 (3) | 5 (12) | 6 (7)
Inpatient psychiatric treatment (Psychiatric disorders) | 1 (2) | 1 (2) | 2 (3) | 1 (1)
Inpatient medical treatment (General disorders) | 2 (2) | 4 (8) | 4 (6) | 4 (5)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A - Standard Job Activity Contracting and Alcohol Monitoring (N=50) | Group B - Reinforcement for Negative Alcohol Samples (N=65) | Group C - Reinforcement for Completing Job Activities (N=58) | Group D - Reinforcement for Negative Alcohol Samples & Job Activities (N=67)
Emergency Room Visit (General disorders) | 5 (6) | 5 (7) | 1 (1) | 6 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-06-15): https://cdn.clinicaltrials.gov/large-docs/09/NCT02559609/Prot_SAP_000.pdf
  • Informed Consent Form (2021-04-29): https://cdn.clinicaltrials.gov/large-docs/09/NCT02559609/ICF_001.pdf